CLINICAL TRIAL: NCT04153708
Title: A Clinical Trial to Evaluate the Efficacy of Two Strategies to Linkage to Care Patients With Hepatitis C Lost to Follow-up
Brief Title: Retrieval of Hepatitis C Patients Lost to Follow-up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of La Laguna (Other)
Responsible Party: Principal Investigator, Manuel Hernandez-Guerra, MD, Principal Investigator, University of La Laguna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUC_2019 23
Record Dates: First submitted 2019-11-03; First posted 2019-11-06 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Hepatitis C
Keywords: hepatitis C; lost to follow-up; microelimination
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to either call or mail invitation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrieval by phone call. (Experimental): Patients assigned to strategy 1 will be called to schedule an appointment with the hepatologist over a period of 14 days.
  Interventions: Behavioral: Retrieval patients lost to follow-up with positive HCV antibodies without RNA request or positive RNA by phone call.
- Retrieval by mail letter (Active Comparator): Patients assigned to strategy 2 will receive an invitation letter with an appointment with the hepatologist over a period of 14 days.
  Interventions: Behavioral: Retrieval patients lost to follow-up with positive HCV antibodies without RNA request or positive RNA by mail letter

INTERVENTIONS:
Behavioral: Retrieval patients lost to follow-up with positive HCV antibodies without RNA request or positive RNA by phone call. — Patients assigned to strategy 1 will be called to schedule an appointment with the hepatologist over a period of 14 days.
  Arms: Retrieval by phone call.
Behavioral: Retrieval patients lost to follow-up with positive HCV antibodies without RNA request or positive RNA by mail letter — Patients assigned to strategy 2 will receive an invitation letter with an appointment with the hepatologist over a period of 14 days.
  Arms: Retrieval by mail letter

SUMMARY:
The main purpose of the study is to compare the efficacy of two strategies aimed to rescue patients lost to follow-up with active infection or with positive HCV antibodies without RNA request to complete evaluation and prescription of treatment in cases of chronic infection. After patient identification from data files of laboratory and microbiology charts, patients will be randomized to: a) phone call, and b) invitation letter, both of two strategies including a scheduled appointment with the hepatologist.

DETAILED DESCRIPTION:
This is a prospective, randomized study in which subjects lost to follow-up with positive HCV antibodies without RNA request or positive RNA will be proposed to be brought back into care.

After patients identification from data files of laboratory and microbiology charts using three different cohorts in time (2005-07, 2011-11 and 2015-17), eligible patients (18 years of age or older, patients positive for HCV antibodies without RNA request or positive RNA lost to follow-up, with a valid sanitary card in our public health system and with available data for contact) will be randomized to: a) phone call (Strategy 1), and b) invitation letter (Strategy 2), both of two strategies including a scheduled appointment with the hepatologist.

Strategy 1 includes until three phone calls to contact patients and provide them with an appointment with the hepatologist (tertiary care center) over a period of 14 days according to patient availability. Instead, strategy 2 includes an invitation letter providing patients with the appointment with the hepatologist over a same period of time than strategy 1. If there is no response to calls or no attendance to the appointment after the letter (randomized strategy), the strategy will be switched to the another one.

Epidemiological, clinical, and laboratory variables will be registered.

The hypothesis of the study is that phone calls will improve the rate of linkage to care among HCV patients lost to follow-up compared to the invitation letter shipment. Therefore, call would be an effective strategy to rescue these patients.

For the present study, a 15% of improvement in linkage to care was hypothesized in the group of patients receiving the strategy 1 compared with the strategy 2. Taking into account a power of 80%, alpha error of 5% and losses of 10% will require 176 patients per strategy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Record of positive HCV antibodies without RNA request or positive RNA lost to follow-up (non-treated patients with an active infection, without surveillance by any HCV specialist)
3. Patients a valid sanitary card in our public health system
4. Patients with available data for contact)

Exclusion Criteria:

1. Belong to another catchment area. Current surveillance by any HCV specialist and/or record of sustained virological response.
2. Severe comorbidity with an expected survival lower than 1 year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 352 (Estimated)
Dates: Start 2019-11-03 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Acceptance of the intervention | One month after the intervention
  Number of patients and % attending the clinic (linkage to care rate)

SECONDARY OUTCOMES:
Effectiveness of the intervention | 6 months after starting treatment
  Number of patients and % that cure the infection due to intervention (complete assessment and treatment rate).
Viability of the intervention | 1 week
  Number of patients with unavailable or inaccurate data for contact
Factors associated with viability of the strategies | 6 months
  Rate of patients with predictive factors associated to outcome 1

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Quintero Carrion, MD, Study Chair — Hospital Universitario de Canarias
Locations (1):
- Manuel Hernandez-Guerra, San Cristóbal de La Laguna, Santa Cruz De Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No